CLINICAL TRIAL: NCT00563381
Title: Effect of Inhalation of Tiotropium Once Daily 18 Mcg Versus Salmeterol Twice Daily 50 Mcg on Time to First Exacerbation in COPD Patients (a Randomised, Double-blind, Double-dummy, Parallel Group, One-year Study).
Brief Title: Tiotropium Once Daily 18 Mcg Versus Salmeterol Twice Daily 50 Mcg on Time to First Exacerbation in COPD Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.389; EUDRACT2007-001840-33
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (2):
- Tiotropium + Placebo (Active Comparator): patients inhale Tiotropium 18mcg once daily via HandiHaler and Placebo MDI twice daily
  Interventions: Drug: Tiotropium bromide; Drug: Placebo Salmeterol
- Salmeterol + Placebo (Active Comparator): patients inhale Salmeterol 50mcg twice daily via MDI and Placebo HandiHaler once daily
  Interventions: Drug: Salmeterol; Drug: Placebo Tiotropium

INTERVENTIONS:
Drug: Tiotropium bromide — 18 mcg/daily
  Arms: Tiotropium + Placebo
Drug: Salmeterol — 100 mcg/daily
  Arms: Salmeterol + Placebo
Drug: Placebo Salmeterol — Placebo identical to Salmeterol device
  Arms: Tiotropium + Placebo
Drug: Placebo Tiotropium — Placebo identical to Tiotropium device
  Arms: Salmeterol + Placebo

SUMMARY:
This is a randomised, double-blind, double-dummy, multinational, multicentre, parallel group trial comparing tiotropium (18 mcg) inhalation capsule via HandiHaler and salmeterol (50 mcg) via MDI in patients with COPD. There will be a two-week run-in period followed by a 52-week randomised treatment phase. Patients who withdraw prematurely from trial medication will be encouraged to remain in the trial and participate in follow-up telephone contacts until their predicted normal exit date from the trial (i.e. 52 weeks after taking the first dose of randomised treatment). The phone calls will be made at all scheduled visits.

The primary objective of this study is to compare the effect of tiotropium (18 mcg) inhalation capsule via HandiHaler with that of salmeterol (50 mcg) via MDI on COPD exacerbations.

The primary endpoint is time to first COPD exacerbation during the 52 week randomised treatment period. A COPD exacerbation will be defined as a complex of respiratory events / symptoms (increase or new onset) of more than one of the following: cough, sputum, wheezing, dyspnoea or chest tightness with at least one symptom lasting at least three days requiring treatment with antibiotics and/or systemic steroids and/or hospitalisation.

The onset of an exacerbation is defined as the onset of the first new or increased reported symptom. The end of the exacerbation should be recorded as defined by the investigator.

Only COPD exacerbations with onset during randomised treatment will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a diagnosis of chronic obstructive pulmonary disease (COPD) and must meet the following criteria at Visit 1:

   Patients must have relatively stable, moderate to very severe airway obstruction with a post-bronchodilator FEV1 <=70% of predicted normal and FEV1 <=70% of FVC post-bronchodilator (i.e. 30 minutes after inhalation of 4 puffs of 100 µg salbutamol or equivalent SABA). Predicted normal values will be calculated according to ECSC.

   For Height measured in inches Males: FEV1 predicted (L) = 4.30 x (height (inches) / 39.37)-0.029 x age (yrs) - 2.49 Females:FEV1 predicted (L) = 3.95 x (height (inches) / 39.37)-0.025 x age (yrs) - 2.60 For Height measured in metres Males: FEV1 predicted (L) = 4.30 x (height (metres)) - 0.029 x age (years) - 2.49 Females: FEV1 predicted (L) = 3.95 x (height (metres)) - 0.025 x age (years) - 2.60
2. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial.
3. Male or female patients 40 years of age or older.
4. Patients with a history of at least one exacerbation within the past year requiring treatment with either antibiotics and/or systemic steroids and/or hospitalisation.
5. Patients must be current or ex-smokers with a smoking history of >= 10 pack-years. (Patients who have never smoked cigarettes must be excluded.)
6. Patients must be able to perform all study-related procedures including technically acceptable pulmonary function tests (PFTs).
7. Patients must be able to inhale medication in a competent manner from the HandiHaler and a metered dose inhaler (MDI).
8. Patients must be able to maintain records (patient daily diary card) during the study period as required in the protocol.

Exclusion Criteria:

1. Significant diseases other than COPD. A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the patients' ability to participate in the study.
2. Patients with a diagnosis of asthma.
3. Patients with a life-threatening pulmonary obstruction, or a history of cystic fibrosis.
4. Patients with known active tuberculosis.
5. Patients with a known symptomatic prostatic hyperplasia or bladder neck obstruction. Patients with symptomatically-controlled prostatic hyperplasia on medication may be included and should continue their medication.
6. Patients with known narrow-angle glaucoma.
7. Patients with a history of myocardial infarction within the year prior to Visit 1.
8. Patients with a history of hospital admission for heart failure within the year prior to Visit 1.
9. Patients with cardiac arrhythmia requiring medical or surgical treatment.
10. Patients with severe cardiovascular disorders.
11. Patients with a known hypersensitivity to anticholinergic drugs, beta-adrenergics, lactose or any other component of the medication delivery system.
12. Patients with known moderate or severe renal insufficiency (known creatinine clearance of <= 50 mL/min).
13. Patients with untreated known hypokalaemia.
14. Patients with untreated known thyrotoxicosis.
15. Patients with brittle/unstable diabetes mellitus.
16. Patients with a history of and/or active significant alcohol or drug abuse. See exclusion criterion 1.
17. Patients who have taken an investigational drug within 30 days or six half-lives (whichever is greater) prior to Screening Visit (Visit 1).
18. Use of systemic corticosteroid medication at unstable doses (i.e less than six weeks on stable dose) or at doses in excess of the equivalent of 10 mg prednisolone per day or 20 mg every other day.
19. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e oral contraceptives, intrauterine devices, diaphragm or subdermal implants e.g Norplant) for at least three months prior to, and for the duration of the trial.
20. Previous participation (receipt of randomised treatment) in this study.
21. Patients who are currently participating in another study.
22. Patients with any respiratory infection or COPD exacerbation in the four weeks prior to the Screening Visit (Visit 1) or during the run-in period should be postponed. In the case of a respiratory infection or COPD exacerbation during the run-in period, the latter may be extended up to four weeks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7376 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (752):
- Austria (18):
  - 205.389.1020 Boehringer Ingelheim Investigational Site, Feldbach
  - 205.389.1010 Boehringer Ingelheim Investigational Site, Feldkirch
  - 205.389.1003 Boehringer Ingelheim Investigational Site, Gänserndorf
  - 205.389.1011 Boehringer Ingelheim Investigational Site, Grimmenstein/Hochegg
  - 205.389.1005 Boehringer Ingelheim Investigational Site, Hallein
  - 205.389.1023 Boehringer Ingelheim Investigational Site, Linz
  - 205.389.1001 Boehringer Ingelheim Investigational Site, Mittersill
  - 205.389.1027 Boehringer Ingelheim Investigational Site, Salzburg
  - 205.389.1026 Boehringer Ingelheim Investigational Site, Schlüsslberg
  - 205.389.1016 Boehringer Ingelheim Investigational Site, Spittal/Drau
  - 205.389.1022 Boehringer Ingelheim Investigational Site, Steyr
  - 205.389.1002 Boehringer Ingelheim Investigational Site, Vienna
  - 205.389.1006 Boehringer Ingelheim Investigational Site, Vienna
  - 205.389.1014 Boehringer Ingelheim Investigational Site, Vienna
  - 205.389.1018 Boehringer Ingelheim Investigational Site, Vienna
  - 205.389.1021 Boehringer Ingelheim Investigational Site, Vienna
  - 205.389.1029 Boehringer Ingelheim Investigational Site, Vienna
  - 205.389.1017 Boehringer Ingelheim Investigational Site, Zwettl Stadt
- Belgium (11):
  - 205.389.1120 Boehringer Ingelheim Investigational Site, Buizingen
  - 205.389.1124 Boehringer Ingelheim Investigational Site, Cerexhe-Heuseux
  - 205.389.1116 Boehringer Ingelheim Investigational Site, Chenée (Liége)
  - 205.389.1121 Boehringer Ingelheim Investigational Site, Dour
  - 205.389.1113 Boehringer Ingelheim Investigational Site, Gembloux
  - 205.389.1117 Boehringer Ingelheim Investigational Site, Gozée
  - 205.389.1126 Boehringer Ingelheim Investigational Site, Hasselt
  - 205.389.1129 Boehringer Ingelheim Investigational Site, Natoye
  - 205.389.1130 Boehringer Ingelheim Investigational Site, Quaregnon
  - 205.389.1115 Boehringer Ingelheim Investigational Site, Thuillies
  - 205.389.1107 Boehringer Ingelheim Investigational Site, Wetteren
- Bulgaria (12):
  - 205.389.3911 Boehringer Ingelheim Investigational Site, Pazardzhik
  - 205.389.3903 Boehringer Ingelheim Investigational Site, Plovdiv
  - 205.389.3915 Boehringer Ingelheim Investigational Site, Plovdiv
  - 205.389.3918 Boehringer Ingelheim Investigational Site, Rousse
  - 205.389.3914 Boehringer Ingelheim Investigational Site, Sliven
  - 205.389.3902 Boehringer Ingelheim Investigational Site, Sofia
  - 205.389.3906 Boehringer Ingelheim Investigational Site, Sofia
  - 205.389.3907 Boehringer Ingelheim Investigational Site, Sofia
  - 205.389.3908 Boehringer Ingelheim Investigational Site, Stara Zagora
  - 205.389.3916 Boehringer Ingelheim Investigational Site, Troyan Municipality
  - 205.389.3912 Boehringer Ingelheim Investigational Site, Varna
  - 205.389.3901 Boehringer Ingelheim Investigational Site, Veliko Tarnovo
- Czechia (29):
  - 205.389.1211 Boehringer Ingelheim Investigational Site, Benešov
  - 205.389.1213 Boehringer Ingelheim Investigational Site, Beroun
  - 205.389.1220 Boehringer Ingelheim Investigational Site, Beroun
  - 205.389.1204 Boehringer Ingelheim Investigational Site, Brno-Královo Pole
  - 205.389.1212 Boehringer Ingelheim Investigational Site, Cheb
  - 205.389.1205 Boehringer Ingelheim Investigational Site, Havlíčkův Brod
  - 205.389.1230 Boehringer Ingelheim Investigational Site, Humpolec
  - 205.389.1208 Boehringer Ingelheim Investigational Site, Jaroměř
  - 205.389.1219 Boehringer Ingelheim Investigational Site, Kyjov
  - 205.389.1225 Boehringer Ingelheim Investigational Site, Liberec
  - 205.389.1218 Boehringer Ingelheim Investigational Site, Litoměřice
  - 205.389.1214 Boehringer Ingelheim Investigational Site, Lovosice
  - 205.389.1207 Boehringer Ingelheim Investigational Site, Neratovice
  - 205.389.1222 Boehringer Ingelheim Investigational Site, Ostrava
  - 205.389.1209 Boehringer Ingelheim Investigational Site, Pilsen
  - 205.389.1216 Boehringer Ingelheim Investigational Site, Pilsen
  - 205.389.1215 Boehringer Ingelheim Investigational Site, Prague
  - 205.389.1217 Boehringer Ingelheim Investigational Site, Prague
  - 205.389.1223 Boehringer Ingelheim Investigational Site, Prague
  - 205.389.1227 Boehringer Ingelheim Investigational Site, Prague
  - 205.389.1229 Boehringer Ingelheim Investigational Site, Prague
  - 205.389.1232 Boehringer Ingelheim Investigational Site, Prague
  - 205.389.1224 Boehringer Ingelheim Investigational Site, Praha 6 - Brevnov
  - 205.389.1228 Boehringer Ingelheim Investigational Site, Přerov
  - 205.389.1231 Boehringer Ingelheim Investigational Site, Rokycany
  - 205.389.1221 Boehringer Ingelheim Investigational Site, Strakonice
  - 205.389.1206 Boehringer Ingelheim Investigational Site, Třemošná
  - 205.389.1210 Boehringer Ingelheim Investigational Site, Znojmo
  - 205.389.1201 Boehringer Ingelheim Investigational Site, Žatec
- Denmark (10):
  - 205.389.1304 Boehringer Ingelheim Investigational Site, Copenhagen
  - 205.389.1301 Boehringer Ingelheim Investigational Site, Elsinore
  - 205.389.1308 Boehringer Ingelheim Investigational Site, Elsinore
  - 205.389.1309 Boehringer Ingelheim Investigational Site, Frederikssund
  - 205.389.1311 Boehringer Ingelheim Investigational Site, Holstebro
  - 205.389.1302 Boehringer Ingelheim Investigational Site, Næstved
  - 205.389.1303 Boehringer Ingelheim Investigational Site, Roskilde
  - 205.389.1310 Boehringer Ingelheim Investigational Site, Skive
  - 205.389.1312 Boehringer Ingelheim Investigational Site, Sønderborg
  - 205.389.1307 Boehringer Ingelheim Investigational Site, Værløse
- Finland (10):
  - 205.389.1402 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.389.1416 Boehringer Ingelheim Investigational Site, Hyvinkää
  - 205.389.1410 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 205.389.1404 Boehringer Ingelheim Investigational Site, Lahti
  - 205.389.1417 Boehringer Ingelheim Investigational Site, Lappeenranta
  - 205.389.1415 Boehringer Ingelheim Investigational Site, Lohja
  - 205.389.1411 Boehringer Ingelheim Investigational Site, Mikkeli
  - 205.389.1409 Boehringer Ingelheim Investigational Site, Pori
  - 205.389.1412 Boehringer Ingelheim Investigational Site, Preitilä Paimio
  - 205.389.1407 Boehringer Ingelheim Investigational Site, Turku
- France (50):
  - 205.389.1607 Boehringer Ingelheim Investigational Site, Baugé
  - 205.389.1525 Boehringer Ingelheim Investigational Site, Beauvais
  - 205.389.1523 Boehringer Ingelheim Investigational Site, Béthune
  - 205.389.1571 Boehringer Ingelheim Investigational Site, Cestas
  - 205.389.1561 Boehringer Ingelheim Investigational Site, Charry Le Rouet
  - 205.389.1507 Boehringer Ingelheim Investigational Site, Cholet
  - 205.389.1554 Boehringer Ingelheim Investigational Site, Ermont
  - 205.389.1606 Boehringer Ingelheim Investigational Site, Écouflant
  - 205.389.1597 Boehringer Ingelheim Investigational Site, La Barre-de-Monts
  - 205.389.1581 Boehringer Ingelheim Investigational Site, La Jubaudière
  - 205.389.1536 Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - 205.389.1598 Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - 205.389.1501 Boehringer Ingelheim Investigational Site, Le Kremlin-Bicêtre
  - 205.389.1503 Boehringer Ingelheim Investigational Site, Le Mans
  - 205.389.1586 Boehringer Ingelheim Investigational Site, Le Pradet
  - 205.389.1528 Boehringer Ingelheim Investigational Site, Marseille
  - 205.389.1530 Boehringer Ingelheim Investigational Site, Marseille
  - 205.389.1558 Boehringer Ingelheim Investigational Site, Marseille
  - 205.389.1564 Boehringer Ingelheim Investigational Site, Marseille
  - 205.389.1565 Boehringer Ingelheim Investigational Site, Marseille
  - 205.389.1539 Boehringer Ingelheim Investigational Site, Montfermeil
  - 205.389.1608 Boehringer Ingelheim Investigational Site, Nantes
  - 205.389.1526 Boehringer Ingelheim Investigational Site, Nice
  - 205.389.1504 Boehringer Ingelheim Investigational Site, Nîmes
  - 205.389.1502 Boehringer Ingelheim Investigational Site, Ollioules
  - 205.389.1541 Boehringer Ingelheim Investigational Site, Orléans
  - 205.389.1527 Boehringer Ingelheim Investigational Site, Perpignan
  - 205.389.1532 Boehringer Ingelheim Investigational Site, Pierre Benite Cédex
  - 205.389.1553 Boehringer Ingelheim Investigational Site, Rennes
  - 205.389.1567 Boehringer Ingelheim Investigational Site, Saint Orens de Cameville
  - 205.389.1555 Boehringer Ingelheim Investigational Site, Saint-Dié
  - 205.389.1514 Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 205.389.1575 Boehringer Ingelheim Investigational Site, Saint-Germain-du-Puch
  - 205.389.1572 Boehringer Ingelheim Investigational Site, Saint-Laurent
  - 205.389.1547 Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
  - 205.389.1577 Boehringer Ingelheim Investigational Site, Saint-Pierre-Montlimart
  - 205.389.1531 Boehringer Ingelheim Investigational Site, Saint-Quentin
  - 205.389.1569 Boehringer Ingelheim Investigational Site, Seysses
  - 205.389.1520 Boehringer Ingelheim Investigational Site, Sélestat
  - 205.389.1510 Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.389.1522 Boehringer Ingelheim Investigational Site, Strasbourg
  - 205.389.1512 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1515 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1519 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1588 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1589 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1590 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1595 Boehringer Ingelheim Investigational Site, Toulon
  - 205.389.1542 Boehringer Ingelheim Investigational Site, Toulouse
  - 205.389.1574 Boehringer Ingelheim Investigational Site, Villenave-d'Ornon
- Germany (164):
  - 205.389.1741 Boehringer Ingelheim Investigational Site, Aachen
  - 205.389.1857 Boehringer Ingelheim Investigational Site, Aalen
  - 205.389.1934 Boehringer Ingelheim Investigational Site, Auerbach
  - 205.389.1868 Boehringer Ingelheim Investigational Site, Augsburg
  - 205.389.1887 Boehringer Ingelheim Investigational Site, Augsburg
  - 205.389.1707 Boehringer Ingelheim Investigational Site, Bad Lippspringe
  - 205.389.1722 Boehringer Ingelheim Investigational Site, Bad Pymont
  - 205.389.1850 Boehringer Ingelheim Investigational Site, Bad Wörishofen
  - 205.389.1765 Boehringer Ingelheim Investigational Site, Bahrdorf
  - 205.389.1792 Boehringer Ingelheim Investigational Site, Beckum
  - 205.389.1801 Boehringer Ingelheim Investigational Site, Bensheim
  - 205.389.1946 Boehringer Ingelheim Investigational Site, Bensheim
  - 205.389.1824 Boehringer Ingelheim Investigational Site, Bergisch Gladbach
  - 205.389.1709 Boehringer Ingelheim Investigational Site, Bergkamen
  - 205.389.1750 Boehringer Ingelheim Investigational Site, Berkatal-Frankershausen
  - 205.389.1701 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1743 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1769 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1789 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1790 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1847 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1855 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1861 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1862 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1867 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1903 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1931 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1932 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1937 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1960 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1969 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1981 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1983 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1984 Boehringer Ingelheim Investigational Site, Berlin
  - 205.389.1747 Boehringer Ingelheim Investigational Site, Bocholt
  - 205.389.1808 Boehringer Ingelheim Investigational Site, Bochum
  - 205.389.1811 Boehringer Ingelheim Investigational Site, Bochum
  - 205.389.1828 Boehringer Ingelheim Investigational Site, Bonn
  - 205.389.1870 Boehringer Ingelheim Investigational Site, Bonn
  - 205.389.1705 Boehringer Ingelheim Investigational Site, Borna
  - 205.389.1809 Boehringer Ingelheim Investigational Site, Brandenburg/Havel
  - 205.389.1859 Boehringer Ingelheim Investigational Site, Bruchsal
  - 205.389.1734 Boehringer Ingelheim Investigational Site, Camburg
  - 205.389.1923 Boehringer Ingelheim Investigational Site, Celle
  - 205.389.1892 Boehringer Ingelheim Investigational Site, Cologne
  - 205.389.1974 Boehringer Ingelheim Investigational Site, Cologne
  - 205.389.1901 Boehringer Ingelheim Investigational Site, Coswig
  - 205.389.1891 Boehringer Ingelheim Investigational Site, Cottbus
  - 205.389.1858 Boehringer Ingelheim Investigational Site, Deggendorf
  - 205.389.1784 Boehringer Ingelheim Investigational Site, Donaueschingen
  - 205.389.1713 Boehringer Ingelheim Investigational Site, Dortmund
  - 205.389.1706 Boehringer Ingelheim Investigational Site, Dresden
  - 205.389.1967 Boehringer Ingelheim Investigational Site, Düren
  - 205.389.1814 Boehringer Ingelheim Investigational Site, Engelskirchen
  - 205.389.1773 Boehringer Ingelheim Investigational Site, Ense
  - 205.389.1727 Boehringer Ingelheim Investigational Site, Eppelborn-Bubach
  - 205.389.1864 Boehringer Ingelheim Investigational Site, Erfurt
  - 205.389.1940 Boehringer Ingelheim Investigational Site, Erlangen
  - 205.389.1900 Boehringer Ingelheim Investigational Site, Eschwege
  - 205.389.1758 Boehringer Ingelheim Investigational Site, Essen
  - 205.389.1975 Boehringer Ingelheim Investigational Site, Essen
  - 205.389.1982 Boehringer Ingelheim Investigational Site, Essen
  - 205.389.1724 Boehringer Ingelheim Investigational Site, Ettlingen
  - 205.389.1806 Boehringer Ingelheim Investigational Site, Feldkirchen-Westerham
  - 205.389.1976 Boehringer Ingelheim Investigational Site, Forchheim
  - 205.389.1943 Boehringer Ingelheim Investigational Site, Föhren
  - 205.389.1795 Boehringer Ingelheim Investigational Site, Frankenberg
  - 205.389.1905 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 205.389.1752 Boehringer Ingelheim Investigational Site, Fuldatal-Ihringshausen
  - 205.389.1971 Boehringer Ingelheim Investigational Site, Fürth
  - 205.389.1766 Boehringer Ingelheim Investigational Site, Gars
  - 205.389.1977 Boehringer Ingelheim Investigational Site, Gelsenkirchen
  - 205.389.1744 Boehringer Ingelheim Investigational Site, Georgensgmünd
  - 205.389.1875 Boehringer Ingelheim Investigational Site, Giessen
  - 205.389.1836 Boehringer Ingelheim Investigational Site, Gifhorn
  - 205.389.1914 Boehringer Ingelheim Investigational Site, Goch
  - 205.389.1751 Boehringer Ingelheim Investigational Site, Göttingen
  - 205.389.1886 Boehringer Ingelheim Investigational Site, Greiz
  - 205.389.1768 Boehringer Ingelheim Investigational Site, Grünberg
  - 205.389.1831 Boehringer Ingelheim Investigational Site, Hagen
  - 205.389.1827 Boehringer Ingelheim Investigational Site, Halle
  - 205.389.1917 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.389.1924 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.389.1925 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.389.1980 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.389.1716 Boehringer Ingelheim Investigational Site, Hammah
  - 205.389.1702 Boehringer Ingelheim Investigational Site, Hammelburg
  - 205.389.1802 Boehringer Ingelheim Investigational Site, Hanover
  - 205.389.1712 Boehringer Ingelheim Investigational Site, Harsewinkel
  - 205.389.1738 Boehringer Ingelheim Investigational Site, Hauzenberg
  - 205.389.1860 Boehringer Ingelheim Investigational Site, Hemmingen
  - 205.389.1949 Boehringer Ingelheim Investigational Site, Höchstädt
  - 205.389.1726 Boehringer Ingelheim Investigational Site, Ingelheim
  - 205.389.1873 Boehringer Ingelheim Investigational Site, Karlsruhe
  - 205.389.1838 Boehringer Ingelheim Investigational Site, Kaufbeuren
  - 205.389.1704 Boehringer Ingelheim Investigational Site, Käbschütztal-Krögis
  - 205.389.1839 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.389.1813 Boehringer Ingelheim Investigational Site, Köthen
  - 205.389.1881 Boehringer Ingelheim Investigational Site, Krefeld
  - 205.389.1786 Boehringer Ingelheim Investigational Site, Krumpa
  - 205.389.1902 Boehringer Ingelheim Investigational Site, Landsberg
  - 205.389.1837 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.389.1841 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.389.1894 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.389.1908 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.389.1874 Boehringer Ingelheim Investigational Site, Leonberg
  - 205.389.1955 Boehringer Ingelheim Investigational Site, Limburg
  - 205.389.1904 Boehringer Ingelheim Investigational Site, Lorch
  - 205.389.1877 Boehringer Ingelheim Investigational Site, Lübeck
  - 205.389.1823 Boehringer Ingelheim Investigational Site, Lützen
  - 205.389.1879 Boehringer Ingelheim Investigational Site, Magdeburg
  - 205.389.1840 Boehringer Ingelheim Investigational Site, Mannheim
  - 205.389.1978 Boehringer Ingelheim Investigational Site, Mannheim
  - 205.389.1866 Boehringer Ingelheim Investigational Site, Marburg
  - 205.389.1871 Boehringer Ingelheim Investigational Site, Marburg
  - 205.389.1926 Boehringer Ingelheim Investigational Site, Marburg
  - 205.389.1776 Boehringer Ingelheim Investigational Site, Marl
  - 205.389.1779 Boehringer Ingelheim Investigational Site, Merrbusch
  - 205.389.1799 Boehringer Ingelheim Investigational Site, München
  - 205.389.1815 Boehringer Ingelheim Investigational Site, München
  - 205.389.1817 Boehringer Ingelheim Investigational Site, München
  - 205.389.1843 Boehringer Ingelheim Investigational Site, München
  - 205.389.1952 Boehringer Ingelheim Investigational Site, Neubrandenburg
  - 205.389.1805 Boehringer Ingelheim Investigational Site, Neuötting
  - 205.389.1948 Boehringer Ingelheim Investigational Site, Neuss
  - 205.389.1958 Boehringer Ingelheim Investigational Site, Neuwied
  - 205.389.1830 Boehringer Ingelheim Investigational Site, Niesky
  - 205.389.1711 Boehringer Ingelheim Investigational Site, Nußbach
  - 205.389.1781 Boehringer Ingelheim Investigational Site, Oberdorla
  - 205.389.1753 Boehringer Ingelheim Investigational Site, Paderborn
  - 205.389.1810 Boehringer Ingelheim Investigational Site, Paderborn
  - 205.389.1854 Boehringer Ingelheim Investigational Site, Paderborn
  - 205.389.1756 Boehringer Ingelheim Investigational Site, Pirmasens
  - 205.389.1794 Boehringer Ingelheim Investigational Site, Potsdam
  - 205.389.1899 Boehringer Ingelheim Investigational Site, Potsdam
  - 205.389.1842 Boehringer Ingelheim Investigational Site, Radebeul
  - 205.389.1897 Boehringer Ingelheim Investigational Site, Rathenow
  - 205.389.1950 Boehringer Ingelheim Investigational Site, Raubach
  - 205.389.1783 Boehringer Ingelheim Investigational Site, Riesa
  - 205.389.1826 Boehringer Ingelheim Investigational Site, Riesa
  - 205.389.1742 Boehringer Ingelheim Investigational Site, Rostock
  - 205.389.1816 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 205.389.1883 Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - 205.389.1878 Boehringer Ingelheim Investigational Site, Saarlouis
  - 205.389.1833 Boehringer Ingelheim Investigational Site, Schmallenberg-Grafschaft
  - 205.389.1973 Boehringer Ingelheim Investigational Site, Schmölln
  - 205.389.1979 Boehringer Ingelheim Investigational Site, Schwetzingen
  - 205.389.1856 Boehringer Ingelheim Investigational Site, Simmern
  - 205.389.1918 Boehringer Ingelheim Investigational Site, Solingen
  - 205.389.1822 Boehringer Ingelheim Investigational Site, Steinfurt
  - 205.389.1728 Boehringer Ingelheim Investigational Site, Sulzbach
  - 205.389.1717 Boehringer Ingelheim Investigational Site, Templin
  - 205.389.1882 Boehringer Ingelheim Investigational Site, Treuenbrietzen
  - 205.389.1745 Boehringer Ingelheim Investigational Site, Wallerfing
  - 205.389.1800 Boehringer Ingelheim Investigational Site, Wardenburg
  - 205.389.1885 Boehringer Ingelheim Investigational Site, Weißenhorn
  - 205.389.1927 Boehringer Ingelheim Investigational Site, Westerstede
  - 205.389.1825 Boehringer Ingelheim Investigational Site, Weyhe
  - 205.389.1863 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 205.389.1968 Boehringer Ingelheim Investigational Site, Wilhelmshaven
  - 205.389.1807 Boehringer Ingelheim Investigational Site, Wilster
  - 205.389.1754 Boehringer Ingelheim Investigational Site, Wolfsburg
  - 205.389.1919 Boehringer Ingelheim Investigational Site, Wuppertal
  - 205.389.1898 Boehringer Ingelheim Investigational Site, Zerbst
- Hungary (29):
  - 205.389.2001 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2005 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2006 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2009 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2016 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2018 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2027 Boehringer Ingelheim Investigational Site, Budapest
  - 205.389.2007 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.389.2035 Boehringer Ingelheim Investigational Site, Deszk
  - 205.389.2015 Boehringer Ingelheim Investigational Site, Dunaújváros
  - 205.389.2008 Boehringer Ingelheim Investigational Site, Érd
  - 205.389.2011 Boehringer Ingelheim Investigational Site, Füzesabony
  - 205.389.2013 Boehringer Ingelheim Investigational Site, Győr
  - 205.389.2028 Boehringer Ingelheim Investigational Site, Gyula
  - 205.389.2014 Boehringer Ingelheim Investigational Site, Jászberény
  - 205.389.2021 Boehringer Ingelheim Investigational Site, Kecskemét
  - 205.389.2025 Boehringer Ingelheim Investigational Site, Komárom
  - 205.389.2024 Boehringer Ingelheim Investigational Site, Mosdós
  - 205.389.2026 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 205.389.2031 Boehringer Ingelheim Investigational Site, Nyíregyháza
  - 205.389.2002 Boehringer Ingelheim Investigational Site, Pécs
  - 205.389.2017 Boehringer Ingelheim Investigational Site, Ráckeve
  - 205.389.2003 Boehringer Ingelheim Investigational Site, Siófok
  - 205.389.2010 Boehringer Ingelheim Investigational Site, Szarvas
  - 205.389.2022 Boehringer Ingelheim Investigational Site, Százhalombatta
  - 205.389.2019 Boehringer Ingelheim Investigational Site, Szentendre
  - 205.389.2030 Boehringer Ingelheim Investigational Site, Tatabánya
  - 205.389.2029 Boehringer Ingelheim Investigational Site, Törökbálint
  - 205.389.2020 Boehringer Ingelheim Investigational Site, Veszprém
- Israel (14):
  - 205.389.2101 Boehringer Ingelheim Investigational Site, Afula
  - 205.389.2110 Boehringer Ingelheim Investigational Site, Ashkelon
  - 205.389.2106 Boehringer Ingelheim Investigational Site, Beersheba
  - 205.389.2112 Boehringer Ingelheim Investigational Site, Hadera
  - 205.389.2107 Boehringer Ingelheim Investigational Site, Haifa
  - 205.389.2111 Boehringer Ingelheim Investigational Site, Haifa
  - 205.389.2108 Boehringer Ingelheim Investigational Site, Holon
  - 205.389.2104 Boehringer Ingelheim Investigational Site, Jerusalem
  - 205.389.2114 Boehringer Ingelheim Investigational Site, Jerusalem
  - 205.389.2116 Boehringer Ingelheim Investigational Site, Nahariya
  - 205.389.2102 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 205.389.2105 Boehringer Ingelheim Investigational Site, Rehovot
  - 205.389.2103 Boehringer Ingelheim Investigational Site, Tel Litwinsky
  - 205.389.2117 Boehringer Ingelheim Investigational Site, Ẕerifin
- Italy (18):
  - 205.389.2211 Boehringer Ingelheim Investigational Site, Brescia
  - 205.389.2206 Boehringer Ingelheim Investigational Site, Cagliari
  - 205.389.2223 Boehringer Ingelheim Investigational Site, Catania
  - 205.389.2209 Boehringer Ingelheim Investigational Site, Ferrara
  - 205.389.2214 Boehringer Ingelheim Investigational Site, Genova
  - 205.389.2215 Boehringer Ingelheim Investigational Site, Lecco
  - 205.389.2221 Boehringer Ingelheim Investigational Site, Milan
  - 205.389.2226 Boehringer Ingelheim Investigational Site, Milan
  - 205.389.2224 Boehringer Ingelheim Investigational Site, Modena
  - 205.389.2203 Boehringer Ingelheim Investigational Site, Montescano (PV)
  - 205.389.2230 Boehringer Ingelheim Investigational Site, Napoli
  - 205.389.2201 Boehringer Ingelheim Investigational Site, Novara
  - 205.389.2229 Boehringer Ingelheim Investigational Site, Pavia
  - 205.389.2227 Boehringer Ingelheim Investigational Site, Pisa
  - 205.389.2205 Boehringer Ingelheim Investigational Site, Roma
  - 205.389.2228 Boehringer Ingelheim Investigational Site, Roma
  - 205.389.2210 Boehringer Ingelheim Investigational Site, Sassari
  - 205.389.2232 Boehringer Ingelheim Investigational Site, Treviso
- Latvia (13):
  - 205.389.2315 Boehringer Ingelheim Investigational Site, Balvi
  - 205.389.2305 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.389.2313 Boehringer Ingelheim Investigational Site, Jelgava
  - 205.389.2311 Boehringer Ingelheim Investigational Site, Krāslava
  - 205.389.2312 Boehringer Ingelheim Investigational Site, Kuldīga
  - 205.389.2301 Boehringer Ingelheim Investigational Site, Riga
  - 205.389.2303 Boehringer Ingelheim Investigational Site, Riga
  - 205.389.2307 Boehringer Ingelheim Investigational Site, Riga
  - 205.389.2310 Boehringer Ingelheim Investigational Site, Riga
  - 205.389.2306 Boehringer Ingelheim Investigational Site, Talsi
  - 205.389.2314 Boehringer Ingelheim Investigational Site, Tukums
  - 205.389.2304 Boehringer Ingelheim Investigational Site, Valmiera
  - 205.389.2302 Boehringer Ingelheim Investigational Site, Ventspils
- Lithuania (14):
  - 205.389.2401 Boehringer Ingelheim Investigational Site, Alytus
  - 205.389.2402 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.389.2403 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.389.2404 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.389.2406 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.389.2409 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.389.2407 Boehringer Ingelheim Investigational Site, Klaipėda
  - 205.389.2411 Boehringer Ingelheim Investigational Site, Klaipėda
  - 205.389.2408 Boehringer Ingelheim Investigational Site, Šiauliai
  - 205.389.2410 Boehringer Ingelheim Investigational Site, Utena
  - 205.389.2405 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.389.2412 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.389.2413 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.389.2414 Boehringer Ingelheim Investigational Site, Vilnius
- Netherlands (4):
  - 205.389.2504 Boehringer Ingelheim Investigational Site, Rotterdam
  - 205.389.2508 Boehringer Ingelheim Investigational Site, Te Leiderdrop
  - 205.389.2510 Boehringer Ingelheim Investigational Site, Velp
  - 205.389.2511 Boehringer Ingelheim Investigational Site, Zoetermeer
- Norway (12):
  - 205.389.2614 Boehringer Ingelheim Investigational Site, Ålesund
  - 205.389.2604 Boehringer Ingelheim Investigational Site, Bekkestua
  - 205.389.2601 Boehringer Ingelheim Investigational Site, Elverum
  - 205.389.2611 Boehringer Ingelheim Investigational Site, Follebu
  - 205.389.2602 Boehringer Ingelheim Investigational Site, Hamar
  - 205.389.2610 Boehringer Ingelheim Investigational Site, Harstad
  - 205.389.2613 Boehringer Ingelheim Investigational Site, Harstad
  - 205.389.2609 Boehringer Ingelheim Investigational Site, Hønefoss
  - 205.389.2608 Boehringer Ingelheim Investigational Site, Lørenskog
  - 205.389.2605 Boehringer Ingelheim Investigational Site, Oslo
  - 205.389.2612 Boehringer Ingelheim Investigational Site, Oslo
  - 205.389.2616 Boehringer Ingelheim Investigational Site, Stavanger
- Poland (93):
  - 205.389.2708 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.389.2744 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.389.2762 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.389.2765 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.389.2778 Boehringer Ingelheim Investigational Site, Bielsko-Biala
  - 205.389.2706 Boehringer Ingelheim Investigational Site, Bieńkówka
  - 205.389.2750 Boehringer Ingelheim Investigational Site, Brzesko
  - 205.389.2758 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 205.389.2773 Boehringer Ingelheim Investigational Site, Bystra
  - 205.389.2800 Boehringer Ingelheim Investigational Site, Chodzież
  - 205.389.2712 Boehringer Ingelheim Investigational Site, Częstochowa
  - 205.389.2774 Boehringer Ingelheim Investigational Site, Częstochowa
  - 205.389.2815 Boehringer Ingelheim Investigational Site, Działdowo
  - 205.389.2787 Boehringer Ingelheim Investigational Site, Elblag
  - 205.389.2715 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.389.2723 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.389.2743 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.389.2764 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.389.2802 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.389.2801 Boehringer Ingelheim Investigational Site, Gorzow Wlkp
  - 205.389.2791 Boehringer Ingelheim Investigational Site, Inowrocław
  - 205.389.2805 Boehringer Ingelheim Investigational Site, Iława
  - 205.389.2705 Boehringer Ingelheim Investigational Site, Katowice
  - 205.389.2749 Boehringer Ingelheim Investigational Site, Katowice
  - 205.389.2771 Boehringer Ingelheim Investigational Site, Katowice
  - 205.389.2759 Boehringer Ingelheim Investigational Site, Koszalin
  - 205.389.2711 Boehringer Ingelheim Investigational Site, Krakow
  - 205.389.2722 Boehringer Ingelheim Investigational Site, Krakow
  - 205.389.2747 Boehringer Ingelheim Investigational Site, Krakow
  - 205.389.2748 Boehringer Ingelheim Investigational Site, Krakow
  - 205.389.2753 Boehringer Ingelheim Investigational Site, Krakow
  - 205.389.2798 Boehringer Ingelheim Investigational Site, Krakow
  - 205.389.2757 Boehringer Ingelheim Investigational Site, Kutno
  - 205.389.2727 Boehringer Ingelheim Investigational Site, Leszno
  - 205.389.2701 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2709 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2716 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2724 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2732 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2746 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2751 Boehringer Ingelheim Investigational Site, Lodz
  - 205.389.2741 Boehringer Ingelheim Investigational Site, Lublin
  - 205.389.2776 Boehringer Ingelheim Investigational Site, Lublin
  - 205.389.2817 Boehringer Ingelheim Investigational Site, Lublin
  - 205.389.2756 Boehringer Ingelheim Investigational Site, Olsztyn
  - 205.389.2816 Boehringer Ingelheim Investigational Site, Olsztyn
  - 205.389.2702 Boehringer Ingelheim Investigational Site, Ostrow Wielkopolska
  - 205.389.2760 Boehringer Ingelheim Investigational Site, Oława
  - 205.389.2726 Boehringer Ingelheim Investigational Site, Pabianice
  - 205.389.2703 Boehringer Ingelheim Investigational Site, Poznan
  - 205.389.2719 Boehringer Ingelheim Investigational Site, Poznan
  - 205.389.2737 Boehringer Ingelheim Investigational Site, Poznan
  - 205.389.2766 Boehringer Ingelheim Investigational Site, Poznan
  - 205.389.2769 Boehringer Ingelheim Investigational Site, Poznan
  - 205.389.2813 Boehringer Ingelheim Investigational Site, Poznan
  - 205.389.2763 Boehringer Ingelheim Investigational Site, Proszowice
  - 205.389.2767 Boehringer Ingelheim Investigational Site, Pruszków
  - 205.389.2795 Boehringer Ingelheim Investigational Site, Pławno
  - 205.389.2730 Boehringer Ingelheim Investigational Site, Płock
  - 205.389.2768 Boehringer Ingelheim Investigational Site, Radom
  - 205.389.2792 Boehringer Ingelheim Investigational Site, Sandomierz
  - 205.389.2781 Boehringer Ingelheim Investigational Site, Sieradz
  - 205.389.2725 Boehringer Ingelheim Investigational Site, Skierniewice
  - 205.389.2718 Boehringer Ingelheim Investigational Site, Szczecin
  - 205.389.2739 Boehringer Ingelheim Investigational Site, Szczecin
  - 205.389.2772 Boehringer Ingelheim Investigational Site, Szczecin
  - 205.389.2777 Boehringer Ingelheim Investigational Site, Szczecin - Zdunowo
  - 205.389.2782 Boehringer Ingelheim Investigational Site, Szczecin - Zdunowo
  - 205.389.2738 Boehringer Ingelheim Investigational Site, Tarnów
  - 205.389.2799 Boehringer Ingelheim Investigational Site, Tarnów
  - 205.389.2810 Boehringer Ingelheim Investigational Site, Tczew
  - 205.389.2775 Boehringer Ingelheim Investigational Site, Torun
  - 205.389.2754 Boehringer Ingelheim Investigational Site, Tranow
  - 205.389.2806 Boehringer Ingelheim Investigational Site, Turek
  - 205.389.2803 Boehringer Ingelheim Investigational Site, Wabrzenzo
  - 205.389.2707 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.389.2714 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.389.2728 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.389.2734 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.389.2812 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.389.2818 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.389.2710 Boehringer Ingelheim Investigational Site, Wodzisław Śląski
  - 205.389.2721 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2731 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2736 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2752 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2761 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2780 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2793 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.389.2783 Boehringer Ingelheim Investigational Site, Zabrze
  - 205.389.2735 Boehringer Ingelheim Investigational Site, Zakopane
  - 205.389.2770 Boehringer Ingelheim Investigational Site, Zgierz
  - 205.389.2804 Boehringer Ingelheim Investigational Site, Łomża
- Portugal (10):
  - 205.389.2912 Boehringer Ingelheim Investigational Site, Angra do Heroísmo
  - 205.389.2911 Boehringer Ingelheim Investigational Site, Barreiro
  - 205.389.2904 Boehringer Ingelheim Investigational Site, Faro
  - 205.389.2910 Boehringer Ingelheim Investigational Site, Figueira da Foz Municipality
  - 205.389.2907 Boehringer Ingelheim Investigational Site, Guarda
  - 205.389.2914 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.389.2917 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.389.2905 Boehringer Ingelheim Investigational Site, Santa Maria da Feira
  - 205.389.2909 Boehringer Ingelheim Investigational Site, Santiago do Cacém
  - 205.389.2903 Boehringer Ingelheim Investigational Site, Torres Vedras
- Romania (21):
  - 205.389.3009 Boehringer Ingelheim Investigational Site, Brasov
  - 205.389.3018 Boehringer Ingelheim Investigational Site, Brasov
  - 205.389.3023 Boehringer Ingelheim Investigational Site, Brasov
  - 205.389.3001 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3002 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3004 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3006 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3007 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3012 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3013 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3025 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.389.3016 Boehringer Ingelheim Investigational Site, Constanța
  - 205.389.3019 Boehringer Ingelheim Investigational Site, Constanța
  - 205.389.3015 Boehringer Ingelheim Investigational Site, Craiova
  - 205.389.3008 Boehringer Ingelheim Investigational Site, Iași
  - 205.389.3014 Boehringer Ingelheim Investigational Site, Iași
  - 205.389.3022 Boehringer Ingelheim Investigational Site, Iași
  - 205.389.3024 Boehringer Ingelheim Investigational Site, Iași
  - 205.389.3005 Boehringer Ingelheim Investigational Site, Oradea
  - 205.389.3017 Boehringer Ingelheim Investigational Site, Tg. Mures
  - 205.389.3021 Boehringer Ingelheim Investigational Site, Timișoara
- Russia (92):
  - 205.389.3174 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 205.389.3113 Boehringer Ingelheim Investigational Site, Barnaul
  - 205.389.3131 Boehringer Ingelheim Investigational Site, Barnaul
  - 205.389.3105 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 205.389.3182 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 205.389.3183 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 205.389.3184 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 205.389.3186 Boehringer Ingelheim Investigational Site, Gatchina (Leningradskaya Oblast)
  - 205.389.3193 Boehringer Ingelheim Investigational Site, Kaliningrad
  - 205.389.3104 Boehringer Ingelheim Investigational Site, Kazan'
  - 205.389.3111 Boehringer Ingelheim Investigational Site, Kemerovo
  - 205.389.3120 Boehringer Ingelheim Investigational Site, Kirov
  - 205.389.3170 Boehringer Ingelheim Investigational Site, Krasnodar
  - 205.389.3132 Boehringer Ingelheim Investigational Site, Krasnoyarsk
  - 205.389.3103 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3106 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3107 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3108 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3109 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3125 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3127 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3128 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3130 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3134 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3136 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3139 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3140 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3143 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3149 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3151 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3156 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3157 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3163 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3164 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3167 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3168 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3171 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3196 Boehringer Ingelheim Investigational Site, Moscow
  - 205.389.3188 Boehringer Ingelheim Investigational Site, Murmansk
  - 205.389.3169 Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - 205.389.3953 Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - 205.389.3112 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.389.3114 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.389.3129 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.389.3141 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.389.3153 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.389.3175 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 205.389.3126 Boehringer Ingelheim Investigational Site, Orenburg
  - 205.389.3185 Boehringer Ingelheim Investigational Site, Perm
  - 205.389.3192 Boehringer Ingelheim Investigational Site, Petrozavodsk
  - 205.389.3179 Boehringer Ingelheim Investigational Site, Pskov
  - 205.389.3190 Boehringer Ingelheim Investigational Site, Pskov
  - 205.389.3199 Boehringer Ingelheim Investigational Site, Pyatigorsk
  - 205.389.3159 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 205.389.3197 Boehringer Ingelheim Investigational Site, Ryazan
  - 205.389.3117 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3119 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3121 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3122 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3123 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3135 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3137 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3145 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3146 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3147 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3152 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3160 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3161 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3176 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3177 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3178 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3180 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3181 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3189 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3191 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3195 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3198 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3950 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.389.3110 Boehringer Ingelheim Investigational Site, Saratov
  - 205.389.3951 Boehringer Ingelheim Investigational Site, Saratov
  - 205.389.3165 Boehringer Ingelheim Investigational Site, St.Peterburg
  - 205.389.3101 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.389.3102 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.389.3133 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.389.3144 Boehringer Ingelheim Investigational Site, Tomsk
  - 205.389.3194 Boehringer Ingelheim Investigational Site, Veliky Novgorod
  - 205.389.3118 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 205.389.3155 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 205.389.3116 Boehringer Ingelheim Investigational Site, Yekaterinburg
  - 205.389.3138 Boehringer Ingelheim Investigational Site, Yekaterinburg
  - 205.389.3148 Boehringer Ingelheim Investigational Site, Yekaterinburg
  - 205.389.3166 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Slovakia (8):
  - 205.389.3208 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.389.3204 Boehringer Ingelheim Investigational Site, Košice
  - 205.389.3209 Boehringer Ingelheim Investigational Site, Košice
  - 205.389.3205 Boehringer Ingelheim Investigational Site, Prievidza
  - 205.389.3210 Boehringer Ingelheim Investigational Site, Revúca
  - 205.389.3203 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
  - 205.389.3202 Boehringer Ingelheim Investigational Site, Trnava
  - 205.389.3207 Boehringer Ingelheim Investigational Site, Vráble
- Slovenia (6):
  - 205.389.3301 Boehringer Ingelheim Investigational Site, Golnik
  - 205.389.3308 Boehringer Ingelheim Investigational Site, Grosuplje
  - 205.389.3304 Boehringer Ingelheim Investigational Site, Jesenice
  - 205.389.3302 Boehringer Ingelheim Investigational Site, Kamnik
  - 205.389.3303 Boehringer Ingelheim Investigational Site, Ljubljana
  - 205.389.3306 Boehringer Ingelheim Investigational Site, Topolšica
- Spain (24):
  - 205.389.3410 Boehringer Ingelheim Investigational Site, Badajoz
  - 205.389.3403 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 205.389.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 205.389.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 205.389.3428 Boehringer Ingelheim Investigational Site, Barcelona
  - 205.389.3430 Boehringer Ingelheim Investigational Site, Cartagena
  - 205.389.3416 Boehringer Ingelheim Investigational Site, Cáceres
  - 205.389.3425 Boehringer Ingelheim Investigational Site, Elche
  - 205.389.3408 Boehringer Ingelheim Investigational Site, Las Palmas de Gran Canarias
  - 205.389.3405 Boehringer Ingelheim Investigational Site, Lleida
  - 205.389.3404 Boehringer Ingelheim Investigational Site, Madrid
  - 205.389.3406 Boehringer Ingelheim Investigational Site, Madrid
  - 205.389.3414 Boehringer Ingelheim Investigational Site, Málaga
  - 205.389.3431 Boehringer Ingelheim Investigational Site, Pontevedra
  - 205.389.3419 Boehringer Ingelheim Investigational Site, Requena
  - 205.389.3427 Boehringer Ingelheim Investigational Site, Reus
  - 205.389.3422 Boehringer Ingelheim Investigational Site, Sagunto
  - 205.389.3420 Boehringer Ingelheim Investigational Site, San Juan
  - 205.389.3415 Boehringer Ingelheim Investigational Site, Santander
  - 205.389.3421 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 205.389.3407 Boehringer Ingelheim Investigational Site, Terrasa (Barcelona)
  - 205.389.3413 Boehringer Ingelheim Investigational Site, Valencia
  - 205.389.3426 Boehringer Ingelheim Investigational Site, Valencia
  - 205.389.3417 Boehringer Ingelheim Investigational Site, Valladolid
- Turkey (Türkiye) (12):
  - 205.389.3821 Boehringer Ingelheim Investigational Site, Adana
  - 205.389.3808 Boehringer Ingelheim Investigational Site, Ankara
  - 205.389.3810 Boehringer Ingelheim Investigational Site, Ankara
  - 205.389.3817 Boehringer Ingelheim Investigational Site, Bursa
  - 205.389.3819 Boehringer Ingelheim Investigational Site, Erzurum
  - 205.389.3812 Boehringer Ingelheim Investigational Site, Istanbul
  - 205.389.3827 Boehringer Ingelheim Investigational Site, Izmir
  - 205.389.3813 Boehringer Ingelheim Investigational Site, İzmit
  - 205.389.3820 Boehringer Ingelheim Investigational Site, Kahramanmaraş
  - 205.389.3825 Boehringer Ingelheim Investigational Site, Malatya
  - 205.389.3809 Boehringer Ingelheim Investigational Site, Sihhiye Ankara
  - 205.389.3807 Boehringer Ingelheim Investigational Site, Yenisehir-IZMIR
- Ukraine (52):
  - 205.389.3521 Boehringer Ingelheim Investigational Site, AR Crimea
  - 205.389.3516 Boehringer Ingelheim Investigational Site, Cherkassy
  - 205.389.3549 Boehringer Ingelheim Investigational Site, Chernivtsi
  - 205.389.3509 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.389.3510 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.389.3511 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.389.3523 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.389.3514 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.389.3524 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.389.3533 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 205.389.3506 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3507 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3508 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3520 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3522 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3532 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3539 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3541 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3543 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3555 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.389.3501 Boehringer Ingelheim Investigational Site, Kiev
  - 205.389.3502 Boehringer Ingelheim Investigational Site, Kiev
  - 205.389.3503 Boehringer Ingelheim Investigational Site, Kiev
  - 205.389.3550 Boehringer Ingelheim Investigational Site, Kiev
  - 205.389.3552 Boehringer Ingelheim Investigational Site, Kiev
  - 205.389.3553 Boehringer Ingelheim Investigational Site, Kiev
  - 205.389.3504 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3525 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3526 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3528 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3534 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3535 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3536 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3538 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3551 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.389.3545 Boehringer Ingelheim Investigational Site, Luhansk
  - 205.389.3512 Boehringer Ingelheim Investigational Site, Lviv
  - 205.389.3530 Boehringer Ingelheim Investigational Site, Lviv
  - 205.389.3540 Boehringer Ingelheim Investigational Site, Lviv
  - 205.389.3554 Boehringer Ingelheim Investigational Site, Lviv
  - 205.389.3556 Boehringer Ingelheim Investigational Site, m.Donetsk
  - 205.389.3513 Boehringer Ingelheim Investigational Site, m.Odesa
  - 205.389.3519 Boehringer Ingelheim Investigational Site, Odesa
  - 205.389.3527 Boehringer Ingelheim Investigational Site, Odesa
  - 205.389.3542 Boehringer Ingelheim Investigational Site, Odesa
  - 205.389.3531 Boehringer Ingelheim Investigational Site, Poltava
  - 205.389.3517 Boehringer Ingelheim Investigational Site, Simferopil
  - 205.389.3518 Boehringer Ingelheim Investigational Site, Ternopil
  - 205.389.3529 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 205.389.3515 Boehringer Ingelheim Investigational Site, Zaporizhzhya
  - 205.389.3547 Boehringer Ingelheim Investigational Site, Zaporizhzhya
  - 205.389.3548 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (26):
  - 205.389.3601 Boehringer Ingelheim Investigational Site, Bath
  - 205.389.3630 Boehringer Ingelheim Investigational Site, Bexhill-on-Sea
  - 205.389.3636 Boehringer Ingelheim Investigational Site, Bexhill-on-Sea
  - 205.389.3608 Boehringer Ingelheim Investigational Site, Birmingham
  - 205.389.3605 Boehringer Ingelheim Investigational Site, Blackburn
  - 205.389.3609 Boehringer Ingelheim Investigational Site, Bolton
  - 205.389.3640 Boehringer Ingelheim Investigational Site, Burbage
  - 205.389.3643 Boehringer Ingelheim Investigational Site, Chesterfield
  - 205.389.3627 Boehringer Ingelheim Investigational Site, Corsham
  - 205.389.3606 Boehringer Ingelheim Investigational Site, Coventry
  - 205.389.3633 Boehringer Ingelheim Investigational Site, Coventry
  - 205.389.3639 Boehringer Ingelheim Investigational Site, Frome
  - 205.389.3602 Boehringer Ingelheim Investigational Site, Glasgow
  - 205.389.3632 Boehringer Ingelheim Investigational Site, Irvine
  - 205.389.3623 Boehringer Ingelheim Investigational Site, London
  - 205.389.3638 Boehringer Ingelheim Investigational Site, Middlesex
  - 205.389.3616 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 205.389.3618 Boehringer Ingelheim Investigational Site, Paisley
  - 205.389.3622 Boehringer Ingelheim Investigational Site, Radstock
  - 205.389.3626 Boehringer Ingelheim Investigational Site, Randalstown
  - 205.389.3613 Boehringer Ingelheim Investigational Site, Saint Just, Penzance
  - 205.389.3604 Boehringer Ingelheim Investigational Site, Soham
  - 205.389.3624 Boehringer Ingelheim Investigational Site, Sunderland
  - 205.389.3635 Boehringer Ingelheim Investigational Site, Wansford, Peterborough
  - 205.389.3631 Boehringer Ingelheim Investigational Site, Windsor
  - 205.389.3612 Boehringer Ingelheim Investigational Site, Wrexham

REFERENCES:
- [Derived] Vogelmeier CF, Asijee GM, Kupas K, Beeh KM. Tiotropium and Salmeterol in COPD Patients at Risk of Exacerbations: A Post Hoc Analysis from POET-COPD((R)). Adv Ther. 2015 Jun;32(6):537-47. doi: 10.1007/s12325-015-0216-2. Epub 2015 Jun 23. PMID 26100349
- [Derived] Rabe KF, Fabbri LM, Israel E, Kogler H, Riemann K, Schmidt H, Glaab T, Vogelmeier CF. Effect of ADRB2 polymorphisms on the efficacy of salmeterol and tiotropium in preventing COPD exacerbations: a prespecified substudy of the POET-COPD trial. Lancet Respir Med. 2014 Jan;2(1):44-53. doi: 10.1016/S2213-2600(13)70248-0. Epub 2013 Dec 5. PMID 24461901
- [Derived] Beeh KM, Glaab T, Stowasser S, Schmidt H, Fabbri LM, Rabe KF, Vogelmeier CF. Characterisation of exacerbation risk and exacerbator phenotypes in the POET-COPD trial. Respir Res. 2013 Oct 29;14(1):116. doi: 10.1186/1465-9921-14-116. PMID 24168767
- [Derived] Rabe KF, Fabbri LM, Vogelmeier C, Kogler H, Schmidt H, Beeh KM, Glaab T. Seasonal distribution of COPD exacerbations in the Prevention of Exacerbations with Tiotropium in COPD trial. Chest. 2013 Mar;143(3):711-719. doi: 10.1378/chest.12-1277. PMID 23188489
- [Derived] Vogelmeier C, Hederer B, Glaab T, Schmidt H, Rutten-van Molken MP, Beeh KM, Rabe KF, Fabbri LM; POET-COPD Investigators. Tiotropium versus salmeterol for the prevention of exacerbations of COPD. N Engl J Med. 2011 Mar 24;364(12):1093-1103. doi: 10.1056/NEJMoa1008378. PMID 21428765
- [Derived] Beeh KM, Hederer B, Glaab T, Muller A, Rutten-van Moelken M, Kesten S, Vogelmeier C. Study design considerations in a large COPD trial comparing effects of tiotropium with salmeterol on exacerbations. Int J Chron Obstruct Pulmon Dis. 2009;4:119-25. Epub 2009 Apr 15. PMID 19436693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 8 patients (4:4 on Tiotropium and Salmeterol respectively) randomized but not treated
Groups:
- Tiotropium: Tiotropium 18 mcg once daily (QD) inhalation (powder) via HandiHaler® and matching Placebo metered dose inhaler (MDI) twice daily (BID)
- Salmeterol: Salmeterol 50 mcg (2 actuations of 25 mcg) twice daily inhalation (suspension) via MDI and Placebo HandiHaler® once daily
Period: Overall Study
Arm/Group | Tiotropium | Salmeterol
Started | 3707 (Started treatment) | 3669 (Started treatment)
Completed | 3122 (Completed treatment) | 3021 (Completed treatment)
Not Completed | 585 | 648
Not completed — Adverse Event | 264 | 292
Not completed — Protocol Violation | 66 | 74
Not completed — Lost to Follow-up | 7 | 15
Not completed — Withdrawal by Subject | 192 | 209
Not completed — Lack of Efficacy | 32 | 24
Not completed — Individual different reasons | 24 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Salmeterol | Total
Number analyzed (Participants) | 3707 | 3669 | 7376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.0) | 62.8 (9.0) | 62.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 948 | 922 | 1870
  Male | 2759 | 2747 | 5506
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 5 | 3 | 8
  Black | 9 | 9 | 18
  White | 3693 | 3657 | 7350

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of (Moderate or Severe) COPD Exacerbation
Description: First occurrence analysed by Cox regression as time to first exacerbation and reported as hazard ratio. An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: All patients who received study medication, were randomised, and were documented to have taken at least one dose of double-blind treatment
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 1277 | 1414
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.83, 95% CI [0.77 to 0.90]

2. Secondary Outcome: COPD Exacerbations Per Patient-year Leading to Hospitalisation
Description: An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Hospitalizations per patient-year
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
Hospitalizations per patient-year | 0.09 [0.09 to 0.10] | 0.13 [0.12 to 0.14]
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium vs. Salmeterol; Test type: Superiority or Other; p < 0.0001, Poisson regression; Poisson regression correcting for overdisperion and adjusted for treatment exposure; Rate ratio (ratio of incidence rates) = 0.73, 95% CI [0.66 to 0.82], Standard Error of Mean 0.04

3. Secondary Outcome: Number of Participants With at Least One COPD Exacerbation
Description: as for outcome 2
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
Participants
  Participants with (at least one) event | 1277 | 1414
  Participants with no event | 2430 | 2255
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.90, 95% CI [0.85 to 0.95]

4. Secondary Outcome: COPD Exacerbations Per Patient-year
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
exacerbations per patient-year | 0.64 [0.61 to 0.67] | 0.72 [0.68 to 0.75]
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0017, Poisson regression; Poisson regression correcting for overdisperion and adjusted for treatment exposure; Rate ratio (ratio of incidence rates) = 0.89, 95% CI [0.83 to 0.96], Standard Error of Mean 0.03

5. Secondary Outcome: First Occurrence of COPD Exacerbation Leading to Hospitalization
Description: First occurrence analysed by Cox regression as time to first exacerbation leading to hospitalisation and reported as hazard ratio. An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 262 | 336
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.72, 95% CI [0.61 to 0.85]

6. Secondary Outcome: Number of Participants With at Least One COPD Exacerbation Leading to Hospitalisation
Description: as for outcome 2
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
Participants
  Participants with (at least one) event | 262 | 336
  Participants with no event | 3445 | 3333
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.77, 95% CI [0.66 to 0.89]

7. Secondary Outcome: Occurrence of Premature Discontinuation of Trial Medication
Description: Occurrence analysed by Cox regression as time to premature discontinuation of trial medication and reported as hazard ratio
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 585 | 648
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0242, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.88, 95% CI [0.78 to 0.98]

8. Secondary Outcome: Number of Participants With Premature Discontinuation of Trial Medication
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
Participants
  Participants with (at least one) event | 585 | 648
  Participants with no event | 3122 | 3021
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0406, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.90, 95% CI [0.82 to 1.00]

9. Secondary Outcome: First Occurrence of COPD Exacerbation or Discontinuation of Trial Medication Because of Worsening of Underlying Disease, Whichever Comes First
Description: First occurrence analysed by Cox regression as time to first exacerbation or discontinuation of trial medication because of worsening of underlying disease, whichever comes first and reported as hazard ratio. An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 1316 | 1448
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.84, 95% CI [0.78 to 0.91]

10. Secondary Outcome: First Occurrence of COPD Exacerbations Treated With Systemic Steroids
Description: First occurrence analysed by Cox regression as time to first exacerbation treated with systemic steroids and reported as hazard ratio. An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 715 | 852
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.77, 95% CI [0.69 to 0.85]

11. Secondary Outcome: First Occurrence of COPD Exacerbations Treated With Antibiotics
Description: First occurrence analysed by Cox regression as time to first exacerbation treated with antibiotics and reported as hazard ratio. An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 1154 | 1259
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.85, 95% CI [0.78 to 0.92]

12. Secondary Outcome: First Occurrence of COPD Exacerbations Treated With Systemic Steroids and Antibiotics
Description: First occurrence analysed by Cox regression as time to first exacerbation treated with systemic steroids and antibiotics and reported as hazard ratio. An exacerbation was defined as an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea, chest tightness), with at least 1 symptom lasting at least 3 days and requiring treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospitalisation (severe exacerbation).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of first occurrences
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
number of first occurrences | 562 | 671
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Treatment effect adjusted for pooled centre; Hazard Ratio (HR) = 0.76, 95% CI [0.68 to 0.86]

13. Secondary Outcome: COPD Exacerbations Treated With Systemic Steroids Per Patient-year
Description: as for outcome 2
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
exacerbations per patient-year | 0.33 [0.31 to 0.36] | 0.41 [0.38 to 0.43]
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Poisson regression; Poisson regression correcting for overdispersion and adjusted for treatment exposure; Rate ratio (ratio of incidence rates) = 0.82, 95% CI [0.76 to 0.90], Standard Error of Mean 0.04

14. Secondary Outcome: COPD Exacerbations Treated With Antibiotics Per Patient-year
Description: as for outcome 2
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
exacerbations per patient-year | 0.53 [0.50 to 0.56] | 0.59 [0.56 to 0.62]
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0036, Poisson regression; Poisson regression correcting for overdisperion and adjusted for treatment exposure; Rate ratio (ratio of incidence rates) = 0.90, 95% CI [0.84 to 0.97], Standard Error of Mean 0.03

15. Secondary Outcome: COPD Exacerbations Treated With Systemic Steroids and Antibiotics Per Patient-year
Description: as for outcome 2
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 3707 | 3669
exacerbations per patient-year | 0.23 [0.21 to 0.24] | 0.28 [0.27 to 0.30]
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p < 0.0001, Poisson regression; Poisson regression correcting for overdisperion and adjusted for treatment exposure; Rate ratio (ratio of incidence rates) = 0.80, 95% CI [0.73 to 0.88], Standard Error of Mean 0.04

16. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 1
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: All patients who received study medication, were randomised, were documented to have taken at least one dose of double-blind treatment, gave informed consent to genotyping, took part in the pre-specified part of the genotyping analysis, and who have evaluable blood samples
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2446 | 2434
liter per minute (L/min) | 222.85 (0.81) | 224.45 (0.81)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.1035, Mixed Effects Repeated Measures Model; Mixed effects repeated measures model (MMRM) (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.60, 95% CI [-3.53 to 0.33]

17. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 2
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2413 | 2377
liter per minute (L/min) | 225.15 (0.81) | 227.21 (0.81)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0369, Mixed Effects Repeated Measures Model; Mixed effects repeated measures model (MRMM)(fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -2.06, 95% CI [-3.99 to -0.12]

18. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 3
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2394 | 2357
liter per minute (L/min) | 226.31 (0.81) | 228.38 (0.81)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0362, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -2.07, 95% CI [-4.00 to -0.13]

19. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 4
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2380 | 2349
liter per minute (L/min) | 227.37 (0.81) | 229.25 (0.81)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.0573, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.88, 95% CI [-3.82 to 0.06]

20. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 5
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2360 | 2335
liter per minute (L/min) | 228.27 (0.81) | 229.37 (0.81)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.2641, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.10, 95% CI [-3.04 to 0.83]

21. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 6
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2351 | 2319
liter per minute (L/min) | 228.80 (0.82) | 229.81 (0.81)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.3068, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.01, 95% CI [-2.95 to 0.93]

22. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 7
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2339 | 2306
liter per minute (L/min) | 229.35 (0.82) | 230.13 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.4299, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.78, 95% CI [-2.72 to 1.16]

23. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 8
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2319 | 2278
liter per minute (L/min) | 229.95 (0.82) | 230.43 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.6277, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.48, 95% CI [-2.42 to 1.46]

24. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 9
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2279 | 2234
liter per minute (L/min) | 229.72 (0.82) | 230.57 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.3931, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.85, 95% CI [-2.80 to 1.10]

25. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 10
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2285 | 2235
liter per minute (L/min) | 230.30 (0.82) | 231.27 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.3297, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.97, 95% CI [-2.92 to 0.98]

26. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 11
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2289 | 2228
liter per minute (L/min) | 230.61 (0.82) | 231.91 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.1904, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.30, 95% CI [-3.25 to 0.65]

27. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 12
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2286 | 2214
liter per minute (L/min) | 231.04 (0.82) | 232.04 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.3172, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.99, 95% CI [-2.94 to 0.95]

28. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 13
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2278 | 2212
liter per minute (L/min) | 231.23 (0.82) | 231.89 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.5017, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.67, 95% CI [-2.62 to 1.28]

29. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 14
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2264 | 2211
liter per minute (L/min) | 231.19 (0.82) | 232.42 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.2174, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.23, 95% CI [-3.18 to 0.72]

30. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 15
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2256 | 2193
liter per minute (L/min) | 231.64 (0.82) | 232.75 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.2682, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -1.10, 95% CI [-3.05 to 0.85]

31. Secondary Outcome: Pre-dose Morning PEFR Measured by Patients at Home During the First Four Months of Randomised Treatment (Weekly Means Will be Calculated), Week 16
Description: PEFR means peak expiratory flow rate and is measured in liter per minute
Time Frame: 16 weeks
Population: as for outcome 16
Measure: Mean (Standard Error); unit: liter per minute (L/min)
Arm/Group | Tiotropium | Salmeterol
Number analyzed (Participants) | 2240 | 2174
liter per minute (L/min) | 232.06 (0.82) | 232.65 (0.82)
Statistical Analysis 1: Comparison: Tiotropium vs Salmeterol; Tiotropium versus Salmeterol; Test type: Superiority or Other; p = 0.5520, Mixed Effects Repeated Measures Model; MMRM (fixed terms: treatment, centre, week, treatment*week; covariates: baseline PEFR, baseline PEFR*week); difference in peak expiratory flow rates = -0.59, 95% CI [-2.55 to 1.36]

ADVERSE EVENTS:
Time Frame: 52 weeks (while on treatment with study drugs + 30 days)
Description: The term "Chronic obstructive pulmonary disease" under "Other Adverse Events" contains number of patients with exacerbations which the investigator entered via AE reporting. They were consolidated with the exacerbation events used for efficacy analysis which were collected via separate designated case report form pages.
Arm/Group | Tiotropium | Salmeterol
Serious Adverse Events (participants affected / at risk) | 545/3707 | 606/3669
Other Adverse Events (participants affected / at risk) | 495/3707 | 581/3669
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=3707) | Salmeterol (N=3669)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Splenitis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 3 | 1
Angina pectoris (Cardiac disorders) | 9 | 5
Angina unstable (Cardiac disorders) | 2 | 2
Arrhythmia (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 12 | 14
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 17 | 21
Cardiac failure acute (Cardiac disorders) | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac fibrillation (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 3 | 0
Cardiopulmonary failure (Cardiac disorders) | 4 | 3
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 4 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 4 | 5
Cor pulmonale chronic (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 4 | 5
Coronary artery insufficiency (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 2 | 1
Dressler's syndrome (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1
Left ventricular failure (Cardiac disorders) | 2 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 20 | 13
Myocardial ischaemia (Cardiac disorders) | 11 | 6
Nodal rhythm (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Postinfarction angina (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 4
Sinoatrial block (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tympanosclerosis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 6 | 3
Eye disorder (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Scleritis (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Anal polyp (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Diverticulitis oesophageal (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 3 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enamel anomaly (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 4 | 6
Chills (General disorders) | 0 | 1
Death (General disorders) | 3 | 7
Device dislocation (General disorders) | 1 | 1
Drowning (General disorders) | 2 | 0
Drug intolerance (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 5 | 0
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 3
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 2 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Actinomycosis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Borrelia infection (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 4 | 3
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 3
Cholangitis suppurative (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Dermatitis infected (Infections and infestations) | 1 | 0
Diabetic gangrene (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Groin abscess (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Lung abscess (Infections and infestations) | 1 | 2
Lyme disease (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 2
Otitis media chronic (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 2
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 54 | 64
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Pyothorax (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 4
Rickettsiosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 5 | 1
Wound sepsis (Infections and infestations) | 1 | 0
Accident at work (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 9 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Frostbite (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 3 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram coronary (Investigations) | 1 | 0
Investigation (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dental alveolar anomaly (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 5
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 7
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to retroperitoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Axonal neuropathy (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 2 | 3
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebral circulatory failure (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 9
Cervical root pain (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 2
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypercapnic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1
Postictal state (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 5 | 2
Transient ischaemic attack (Nervous system disorders) | 3 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 3
Drug abuse (Psychiatric disorders) | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 4 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Allergic granulomatous angiitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 270 | 335
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Social problem (Social circumstances) | 1 | 0
Alcohol detoxification (Surgical and medical procedures) | 0 | 1
Intraocular lens implant (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 0
Vocal cord polypectomy (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 2 | 4
Aortic dissection (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 3 | 3
Arteriosclerosis obliterans (Vascular disorders) | 1 | 2
Arteriovenous fistula (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 5 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 1
Embolism (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 9 | 5
Hypertensive crisis (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 1 | 0
Vascular occlusion (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=3707) | Salmeterol (N=3669)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 495 | 581

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.